CLINICAL TRIAL: NCT03810742
Title: Phase 1 Study of Nanoliposomal Irinotecan (Nal-IRI, ONIVYDE®) in Combination With TAS-102 (LONSURF®) in Refractory Solid Tumors
Brief Title: Nanoliposomal Irinotecan (Nal-IRI, ONIVYDE®) in Combination With TAS-102 (LONSURF®) in Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP0210
Record Dates: First submitted 2018-12-21; First posted 2019-01-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Refractory Solid Tumors
MeSH Terms: interventions — irinotecan sucrosofate; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanoliposomal Irinotecan + TAS-102 (Experimental): different dosage combination by Nanoliposomal Irinotecan (nal-IRI, ONIVYDE®) in Combination with TAS-102 (LONSURF®)
  Interventions: Drug: Nanoliposomal Irinotecan

INTERVENTIONS:
Drug: Nanoliposomal Irinotecan — Nanoliposomal Irinotecan (nal-IRI, ONIVYDE®) in Combination with TAS-102 (LONSURF®)
  Other Names: TAS-102

SUMMARY:
The study is to explore the combination of nal-IRI and TAS-102, which is expected to be an effective regimen that could be applied to various cancers

DETAILED DESCRIPTION:
Primary Objectives

* to determine the maximum tolerated dose (MTD) of nal-IRI (ONIVYDE®) in combination with TAS-102 (LONSURF®)
* to evaluate the toxicity profile of the combination therapy Secondary Objectives
* to evaluate the preliminary efficacy of the combination therapy of nal-IRI (ONIVYDE®) and TAS-102 (LONSURF®)
* to study the pharmacokinetics of the combination therapy

A phase 1 study with a classical 3 + 3 dose escalation design. The target population is patients who have pathologically confirmed malignant solid tumors with no standard treatment available.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 20 to 70 years old
2. Histologically or cytologically confirmed malignant solid tumors which are advanced or metastatic, have failed standard treatment or have no standard treatment currently available
3. ECOG performance status 0 or 1
4. Normal ECG or ECG without any clinically significant findings
5. Adequate hematologic parameters, and hepatic and renal function i. White blood cell (WBC) count 3000/μL and absolute neutrophil count (ANC) 1500/μL ii. Platelet counts 100,000/μL without platelet transfusion within 14 days iii. Hemoglobin level 10 g/dL iv. Serum total bilirubin- within normal range v. Serum albumin 3.0 g/dL vi. Serum alanine aminotransferase (ALT) 3 x the upper limit of normal (ULN) vii. Serum creatinine 1.5 x ULN

Exclusion Criteria:

1. Received prior nal-IRI (ONIVYDE®) or TAS-102 (LONSURF®) therapy
2. Known hypersensitivity to any of the components of nal-IRI, other liposomal products, fluoropyrimidines or leucovorin
3. Have liver cirrhosis with Child-Pugh B or Child-Pugh C
4. With active CNS metastasis (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive growth)
5. With clinically significant gastrointestinal disorder including hepatic disorders, bleeding, inflammation, occlusion, or diarrhea > grade 1
6. Life expectancy of less than 3 months
7. Use any anti-cancer or investigational product within 14 days prior to the first date of study dosing
8. History of any second malignancy in the latest 5 years except curatively treated non-melanoma skin cancer or treated cervical carcinoma in situ
9. Uncontrolled inter-current illness including, but not limited to, ongoing or active infection requiring antibiotic treatment, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia, and psychiatric illness or social situation that would preclude study compliance
10. Homozygous for the UGT1A1 28 allele (TA7/TA7), homozygous for UGT1A1 6 allele (A/A), or double heterozygous for both UGT1A1 28 allele (TA6/TA7) and UGT1A1 6 allele (G/A) (only for dose-finding phase)
11. Pregnant or breastfeeding women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Determination of Dose Limiting Toxicities (DLT) | 12 months
  to find the Dose Limiting Toxicity (DLT) of nal-IRI (ONIVYDE®) in combination with TAS-102 (LONSURF®)
Evaluation of Safety profile of nal-IRI and TAS-102 - Incidence of Treatment-Emergent Adverse Events | 12 months
  Incidence of Treatment-Emergent Adverse Events [Safety] of nal-IRI (ONIVYDE®) in combination with TAS-102 (LONSURF®) according to NCI-CTCAE version 5.0

SECONDARY OUTCOMES:
Evaluation of objective tumor response as per Response Evaluation Criteria in Solid Tumors (RECIST) | 24 months
  the objective tumor rate by using RECIST v1.1
Pharmacokinetics study - (Cmax) | 6 months
  Concentration of Peak Plasma (Cmax)
Pharmacokinetics study - (Tmax) | 6 months
  maximum concentration of the time taken to reach the (Tmax).
Pharmacokinetics study - (T1/2) | 6 months
  time of C max to drop in half taken (T1/2)
Pharmacokinetics study - (AUC0→t) | 6 months
  area of the plasma concentration versus time curve (AUC0→t).
Pharmacokinetics study - (AUC0→∞) | 6 months
  area of the plasma concentration versus under curve (AUC0→∞)
Pharmacokinetics study - (CL) | 6 months
  rate of clearance (CL)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chi Lin, MD, Principal Investigator — National Taiwan University Hospital, Taipei, Taiwan
Locations (2):
- Taiwan (2):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan

IPD SHARING:
Plan to Share IPD: No